CLINICAL TRIAL: NCT04639713
Title: A Prospective, Multicenter, Single-Arm Clinical Study Evaluating the Safety and Effectiveness of The Tixel Fractional System in The Treatment of Periorbital Wrinkles
Brief Title: Clinical Study Evaluating the Safety and Effectiveness of The Tixel Fractional System in The Treatment of Periorbital Wrinkles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Novoxel Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN 0749
Record Dates: First submitted 2020-11-19; First posted 2020-11-20 (Actual); Results first posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-02

CONDITIONS: Wrinkle; Periorbital; Tixel 2; Fractional; Resurfacing

STUDY DESIGN:
Intervention Model Description: All participants will undergo treatment with Tixel 2 Device - 4 treatments, 4 weeks apart and 2 Follow Up visits
Masking Description: Blinded assessed of the improvement would be done between Last FU images and baseline, following randomization of the images.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Tixel 2 (Experimental): Tixel 2 Treatment, 4 treatment sessions, followed by 2 Follow up sessions, 1and 3 months after last treatment visit. Subject would be questioned about pain level, subjective dountime assessment and subjective response assessment. Images would be taken at baseline and in Follow-Up visits
  Interventions: Device: Tixel 2

INTERVENTIONS:
Device: Tixel 2 — Thermo-mechanical technology for fractional treatment of human skin. Dermal heating and coagulative effect that occur during the treatment session provide dermal remodeling and collagen restructuring that promote wrinkles appearance improvement.

SUMMARY:
A Prospective, Multicenter, Single-Arm Clinical Study of 51 study subjects who are seeking a procedure to reduce the appearance of the peri-orbital wrinkles. Up to 5 investigational centers in Israel and the United States will participate in the recruitment. Each study subject will receive four (4) treatments with Tixel in a monthly interval. Follow-up will occur 1 month and 3 months following last treatment.

DETAILED DESCRIPTION:
A Prospective, Multicenter, Single-Arm Clinical Study of 51 subjects who are seeking a procedure to reduce the appearance of the periorbital wrinkles, and meet study eligibility criteria, and have provided informed consent will be enrolled in the study. Up to 5 investigational centers in Israel and the United States will participate in the recruitment. Each study subject will receive 4 treatments with Tixel in a monthly interval. Follow-up will occur at 1 month and 3 months following the last treatment.

The clinic visits will be as follow:

1. Baseline (1st tx)
2. Phone-call visit (3 days after the first treatment)
3. 4wk (2nd tx)
4. 8wk (3rd tx)
5. 12wk (4th tx)
6. 4 weeks after the last treatment (1st FU)
7. 12 weeks after the last treatment (2nd FU= 3 months FU, primary endpoint and study completion visit) Primary Efficacy Endpoint is the comparison of the proportion of subjects with a ≥ 1-score improvement on the FWCS at the 3-month visit compared to baseline as determined by at least 2 out of 3 blinded Independent Photographic Reviewers.

Primary Safety Endpoint is the evaluation of related adverse events up to the 3-month visit after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 35-70 years old diagnosed with clinically evident fine (mild) to moderate depth periorbital wrinkling
2. Willingness and ability to comply with all required study activities including returning for follow-up visits and protocol requirements.
3. The subject is able to provide written informed consent and perform the study's activities according to HIPAA guidelines and/or Israeli law, depending on each specific study site.
4. Fitzpatrick wrinkle score of 3-7 in the peri-orbital areas per the treating investigator and clinically noticeable wrinkles in the treating area.
5. Stable body weight during the study period.
6. Skin Type I - V as per Fitzpatrick Skin Scale

Exclusion Criteria:

1. Past treatment with Tixel device.
2. The subject may not undergo treatment by the Tixel device according to the device's contra-indications for use, as defined in the User Manual and in the Instructions for Use and by any other labeling of the device.
3. Subjects who, in the investigator's opinion, have a history of poor cooperation, noncompliance with medical treatment, or unreliability.
4. Female subjects who are pregnant, or planning to become pregnant, or have given birth less than 3 months ago or are lactating.
5. Subjects with significant exposure to critical amounts of ultraviolet light (Sun-tan).
6. Subjects who have had the following treatments:

   1. a cosmetic procedure to improve peri-orbital rhytides (i.e. periorbital or eyelid/eyebrow surgery, brow lift, CO2/Erbium/similar laser/fractional resurfacing, radiofrequency treatment) within 12 months
   2. prior facial treatments with laser, surgical, chemical or light-based facial treatments within the previous 12 months, over the periorbital area including botulinum toxin injections, microdermabrasion or prescription level glycolic acid treatments.
   3. Injectable filler in cheeks (mid face) temples and in the upper face area to be treated within 12 months of investigation.
7. Any subject who have visible scars or other visible changes over the treated areas that may affect evaluation of response and/or quality of photography.
8. Subjects with any type of active cut, wound, inflammation, lesion (benign, premalignant or malignant) or active bacterial, viral, fungal, or herpetic infection on the skin on the designated treatment sites or in close proximity to it.
9. Existing or history of the following (when discussing skin conditions, refers only to the periorbital sites):

   1. skin malignancy, or any diagnosis of suspected malignancy
   2. Collagen or vascular or bleeding disease
   3. Immunosuppression or autoimmune disease
   4. Erythema with or without blistering
   5. History of post inflammatory hyperpigmentation.
   6. Active Acne Vulgaris, HSV-1, or any existing skin condition/disease that in the investigator's opinion would interfere with the evaluation of the safety of the study treatment and evaluation.
   7. Any skin pathology which can induce bullous lesions, urticaria, or demonstrate a Koebner phenomenon (psoriasis, lichen planus, etc.).
   8. Any disease that inhibits pain sensation
   9. History of keloid formation, or hypertrophic scarring
   10. Conditions affecting healing rate (i.e. diabetes mellitus I or II, vascular condition, etc.)
   11. neuromuscular disorders
10. Subjects who have used, within 30 days, any medication that can cause dermal hypersensitivity or affect skin characteristics over the treated area (i.e. topically applied Retinoids, Hydroquinone, Chemical peel of any strength: glycolic acid, lactic acid, salicylic acid)
11. Subjects who have used, systemic treatment which may induce dyspigmentation, such as amiodarone, clofazinmine, minocycline or chloroquine.
12. Subjects currently taking or have taken an oral retinoid in the past six months; Subjects currently taking long-term oral steroid treatment.
13. Concurrent therapy that, in the principal investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study treatment.
14. Subjects who anticipate the need for major surgery or overnight hospitalization during the study that can affect the study schedule or treatment evaluation.
15. Enrollment in any active study involving the use of investigational devices or drugs.
16. Any other cause per the principal investigator's discretion.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerome M Garden, MD, Principal Investigator — Physicians Laser and Dermatology Institute
Locations (3):
- United States (2):
  - Physicians Laser and Dermatology Institute, Chicago, Illinois
  - Laser & Skin Surgery Center of New York, New York, New York
- Rabin Medical Center, Ha'Sharon Campus, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tixel 2
Started | 51
Completed | 48
Not Completed | 3
Not completed — Protocol Noncompliance | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Tixel 2
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (7.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 49
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 15
  Israel | 36

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Safety Adverse Events
Description: Evaluation of related adverse events up to the 3-month after a treatment visit.
Time Frame: 6 months
Measure: Number; unit: Percentage of Participants
Arm/Group | Tixel 2
Number analyzed (Participants) | 51
Percentage of Participants | 3.92

2. Primary Outcome: The Mean Improvement and Treatment Effectiveness by Blinded Assessors Using Using the Fitzpatrick Wrinkle Classification Scale (FWCS) Evaluation
Description: Comparison of the proportion of subjects with a ≥ 1-score improvement on the Fitzpatrick Wrinkle Classification Scale (FWCS) at the 3-month visit compared to baseline as determined by at least 2 out of 3 blinded Independent Photographic Reviewers. The FWCS is a clinically validated assessment tool used to assess skin wrinkle severity and elastosis on a scale from 1 through 9, where the lower score is considered better.
Time Frame: baseline and at 3 months
Population: subjects who received at least one tixel treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Tixel 2: Tixel 2 Treatment, 4 treatment sessions, followed by 2 Follow up sessions, 1 and 3 months after last treatment visit. Subject would be questioned about pain level, subjective downtime assessment and subjective response assessment. Images would be taken at baseline and in Follow-Up visits
  Tixel 2: Thermo-mechanical technology for fractional treatment of human skin. Dermal heating and coagulative effect that occur during the treatment session provide dermal remodeling and collagen restructuring that promote wrinkles appearance improvement.
Arm/Group | Tixel 2
Number analyzed (Participants) | 48
score on a scale
  Assessed by evaluator #1 | 2.00 (0.83)
  Assessed by evaluator #2 | 2.17 (0.71)
  Assessed by evaluator #3 | 1.19 (0.55)

3. Secondary Outcome: The Mean Evaluation of Improvement Assessed by the Handling Physician by Using GAIS Scale - Global Aesthetic Improvement Scale Assessment
Description: Assessment of improvement using Global Aesthetic Improvement Scale Assessment at each visit compared to baseline by the handling physician. Rating:
  1) expectational improvement; 2) very improved patient; 3) Improved patient; 4) Unaltered patient; 5) Worsened patient
Time Frame: Baseline and 3 months visits
Population: subjects who received Tixel treatments
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tixel 2
Number analyzed (Participants) | 48
score on a scale
  GAIS at visit 5 - 1 month FU | 3.54 (0.68)
  GAIS at visit 6 - 3 months FU | 3.52 (0.58)

4. Secondary Outcome: The Mean Score Evaluation of the Pain and Discomfort for Each Treatment
Description: Evaluation of the pain and discomfort of the treatment as reported by the subject on a visual analog scale (VAS). Scoring will consist of making a mark on a 10-points scale. Each line will be awarded a score of 0 - 10 according to the level of pain when 0 is no pain and 10 is the maximum pain possible.
Time Frame: Up to 6 months
Population: pain and discomfort following treatment, reported by the subjects who treated with tixel
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tixel 2
Number analyzed (Participants) | 51
score on a scale
  procedure-associated VAS - treatment 1 | 2.98 (1.52)
  procedure-associated VAS - treatment 2: number analyzed (Participants) | 49
  procedure-associated VAS - treatment 2 | 2.94 (1.14)
  procedure-associated VAS - treatment 3: number analyzed (Participants) | 49
  procedure-associated VAS - treatment 3 | 2.82 (1.22)
  procedure-associated VAS - treatment 4: number analyzed (Participants) | 48
  procedure-associated VAS - treatment 4 | 2.81 (1.2)

5. Secondary Outcome: Satisfaction Questionnaire
Description: Subject Experience (Satisfaction) questionnaire - Subjects assessed their satisfaction at the follow up visits. The following parameters were assessed: results of treatment, treatment experience and expectations (indicating whether the treatment has fulfilled the subject's expectations). For each parameter, the assessment was based on a 5-point scale: 1 = "Poor - Poor or not satisfied at all", 2 ="Fair - satisfied to some extent", 3 = "Moderately - Satisfied", 4 = "Good - Satisfied", 5 = "Excellent - Very Satisfied".
Time Frame: up to 6 months
Population: subject who treated with tixel
Measure: Count of Participants; unit: Participants
Arm/Group | Tixel 2
Number analyzed (Participants) | 48
Participants
  'Very satisfied' with the results of the treatment | 23
  'Very satisfied' with the treatment experience | 33
  'Very satisfied' with regard to their expectations from treatment | 21

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Tixel 2
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 2/51
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tixel 2 (N=51)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) — Erythema
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Back pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-04): https://cdn.clinicaltrials.gov/large-docs/13/NCT04639713/Prot_SAP_000.pdf